CLINICAL TRIAL: NCT02563392
Title: Does Preventive Uterine Artery Occlusion During Laparoscopic Myomectomy Impact on Ovarian Reserve Markers? A Randomized Control Trial
Brief Title: Does Preventive Uterine Artery Occlusion During Laparoscopic Myomectomy Impact on Ovarian Reserve Markers?
Acronym: ORAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Isabelle Streuli, Dr, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-129
Record Dates: First submitted 2015-07-09; First posted 2015-09-30 (Estimated); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Uterine Myoma
MeSH Terms: conditions — Myofibroma | interventions — Uterine Myomectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uterine arteries occlusion (Experimental): Laparoscopic myomectomy with preventive uterine arteries occlusion
  Interventions: Procedure: uterine myomectomy with preventive uterine arteries occlusion
- No uterine arteries occlusion (Active Comparator): Laparoscopic myomectomy without preventive uterine arteries occlusion
  Interventions: Procedure: laparoscopic uterine myomectomy without preventive uterine arteries occlusion

INTERVENTIONS:
Procedure: uterine myomectomy with preventive uterine arteries occlusion — laparoscopic uterine myomectomy with preventive uterine arteries occlusion
  Arms: Uterine arteries occlusion
Procedure: laparoscopic uterine myomectomy without preventive uterine arteries occlusion — laparoscopic uterine myomectomy
  Arms: No uterine arteries occlusion

SUMMARY:
Hysterectomy is an effective treatment used as a first-line approach for uterine myomas. Several others alternatives to hysterectomy have been developed in recent years for women wishing to retain their uterus: myomectomy, radiological embolization, focused ultrasound.

Myomectomy, particularly through minimally invasive surgery, is currently considered the conservative treatment of choice for patients wishing to preserve their fertility. However, three important issues should be considered: the risk of intra- and postoperative bleeding, the risk for recurring myomas, and the preservation of subsequent fertility.

Preventive uterine artery occlusion can be combined with laparoscopic myomectomy in order to avoid bleeding and improve uterine suture. Another expected long-term benefit is the improvement of treatment efficacy, leading to less symptoms and myomas recurrence. However, the effect of uterine arteries occlusion on the ovarian reserve of women of childbearing age has not yet been studied, which limits its clinical application.

DETAILED DESCRIPTION:
Objectives:

1. To assess the effect of preventive uterine artery occlusion during laparoscopic myomectomy on ovarian reserve parameters;
2. To evaluate the effect of preventive uterine artery occlusion during laparoscopic myomectomy on intra- and postoperative blood loss, operative time, clinical symptoms improvement, long-term recurrence of myomas and fertility.

Materials and methods:

Design: This is a prospective randomized single blind trial, including 60 women undergoing a laparoscopic myomectomy for symptomatic uterine myomas. Patients are randomized into two groups: a control group "myomectomy alone" and an experimental group "myomectomy with preventive uterine arteries occlusion".

Setting: The duration of the study will normally be 5 years and will take place at the University Hospitals of Geneva. The study will include about 20 women per year and follow-up will last 2 years. Inclusion criteria are: women of childbearing age, wishing to retain their uterus, having symptomatic uterine myomas and who are eligible for a laparoscopic myomectomy.

The parameters that will be intraoperatively evaluated are the operation time, blood loss and the complications of the surgical technique. Postoperative complications, improving clinical symptoms, myomas recurrence and fertility are discussed at short and long term follow-up.

The ovarian reserve will be evaluated pre- and postoperatively for each patient. It will be determined by plasmatic AMH (anti-Mullerian Hormone) and ultrasound antral follicle count. Women with undetectable preoperative plasmatic AMH will be excluded from the study. Plasmatic AMH and antral follicle count will be measured at 1, 3, 6, 12 and 24 months during the postoperative follow-up.

Limitations:

The sample size is calculated in order to demonstrate a significant difference in plasmatic AMH before and after myomectomy. Small differences are not highlighted in this study, but they probably would not have any impact in clinical practice.

Impact of the study:

The results of this study could have a real impact on daily surgical practice. In case of persistent alteration of ovarian reserve in the experimental group compared to the control group, preventive uterine arteries occlusion during a laparoscopic myomectomy should only be indicated in patients who do not wish pregnancy. If there is no significant impact on ovarian reserve and a beneficial effect on reducing intraoperative blood loss and long-term improvement of symptoms, it should be systematically proposed in all patients undergoing a laparoscopic myomectomy.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* signed the surgery consent form
* capable of discernment understanding and accepting the risks and benefits of the operation
* symptomatic : menorrhagia, breakthrough bleeding and / or pelvic pain and / or infertility and / or repeated spontaneous abortions.
* uterine myoma or more, including at least one type of myoma FIGO 2-6 (International Federation of Gynecology and Obstetrics) objectified by ultrasound and / or pelvic MRI
* laparoscopic approach is technically feasible (as recommended by the National College of Obstetrics and Gynecology French published in 2011): myoma single lower or equal to 9 cm or sum of the size of myomas in centimeters or less equal to 13 and number of myomas inferior to four.
* Female patients of childbearing age younger than 45 years and having a plasma AMH (anti-Mullerian hormone) than 3 pmol / l.
* Patients who accept a postoperative follow-up of 2 years

Exclusion Criteria:

* pregnant patients.
* who underwent radiological uterine artery embolization.
* who have an undetectable AMH levels (<3 pmol / l).
* over 45 years

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2024-05 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
Evolution of ovarian reserve markers after myomectomy | Evaluation of the ovarian reserve at several times: on preoperative, 1, 3, 6, 12 and 24 months postoperative
  It will be determined by plasmatic AMH and ultrasound antral follicle count

SECONDARY OUTCOMES:
Intra-and post-operative blood loss | peroperative
  Blood loss will be estimated during the operation, and will be followed for the duration of hospital stay, an expected average of 3 days. furthermore, we will dose the hemoglobin before and after the intervention.
operative time | peroperative
  Time needed to realise the intervention from the incision to the cutaneous stitches
peroperative complications | peroperative
  it will be noticed the conversion in laparotomy, the blood transfusion, the organic and vessels lesions
Clinical symptoms improvement: hypermenorrhea | 1, 3, 6, 12 and 24 months postoperative
  Evaluation of quantity of blood during menstruation with the PBAC scale (Pictorial Blood Assessment Chart) before and after the intervention
Clinical symptoms improvement: dysmenorrhea | 1, 3, 6, 12 and 24 months postoperative
  Evaluation of improvement of dysmenorrhea by asking patients the pain they have from 0 to 10 and their consumption of pain killers (NSAIDs and paracetamol) during menstruation.
Clinical symptoms improvement: occuring of pregnancy | 12 and 24 months postoperative
  Evaluation of the occurence of pregnancy by asking women the number of pregnancy, of miscarriage, of abortion, of term pregnancy since the intervention
long-term recurrence of myomas | 2 years
  An US will be made at 1, 3, 6, 12 and 24 months to estimate the recidive of myoma. It will be considered a recidive when the myoma will be bigger than 20 mm

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Petignat, Pr, Study Director — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Service de gynécologie, Geneva, Switzerland

REFERENCES:
- [Derived] Streuli I, Ramyead L, Silvestrini N, Petignat P, Dubuisson J. Impact of definitive uterine artery occlusion on ovarian reserve markers in laparoscopic myomectomy: a randomized controlled trial with 2-year follow-up. Hum Reprod. 2025 Jul 1;40(7):1305-1314. doi: 10.1093/humrep/deaf070. PMID 40420404